CLINICAL TRIAL: NCT03243942
Title: Noninvasive, Subharmonic Intra-Cardiac Pressure Measurement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: American Heart Association (Other); Lantheus Medical Imaging (Industry)
Responsible Party: Principal Investigator, Jaydev Dave, Assistant Professor, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15SDG25740015
Record Dates: First submitted 2017-08-03; First posted 2017-08-09 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Cardiac Catheterization; Blood Pressure; Heart Ventricles; Echocardiography; Heart Failure
Keywords: pressure measurements; blood pressure; contrast echocardiography; ventricular pressures; catheterization
MeSH Terms: conditions — Heart Failure | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Definity for pressure measurements (Experimental): 2 vials of activated Definity mixed with 50 ml saline. As per manufacturer's recommendation the infusion rate may vary between 4-10 ml/min (to provide diagnostic intracardiac contrast visibility).
  Interventions: Drug: Definity

INTERVENTIONS:
Drug: Definity — Whenever a patient undergoes cardiac catheterization, which routinely includes intracardiac pressure monitoring using a pressure catheter, as part of their standard clinical care and agrees to participate in the study, we will acquire research data. With Definity infusion, SHAPE algorithm will be initiated to determine optimum acoustic pressure. Then, at the optimum acoustic pressure SHAPE specific data will be acquired from the cardiac chambers and aorta synchronously with the pressures recorded by the catheter (as a part of the patient's standard of care). After acquiring the ultrasound imaging data, the remainder of the heart catheterization will be completed by the attending cardiologist according to the patients' standard of care.

SUMMARY:
The fundamental hypothesis of this project is that real-time intracardiac pressures can be monitored and quantified noninvasively in humans using a novel contrast-enhanced ultrasound technique called subharmonic-aided pressure estimation (SHAPE).This study will use contrast echocardiography to assess the accuracy of SHAPE compared to simultaneously acquired intracardiac pressures measured invasively during cardiac catheterization. This study is designed to verify that contrast echocardiography using the SHAPE method, already proven in a canine model and tested in a human pilot study can be used as a surrogate for cardiac catheterization with sufficient accuracy to allow clinical applicability in humans.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled for a cardiac catheterization procedure
* Adult patients over the age of 21
* Acceptable baseline echocardiographic images in the supine position
* If a female of child-bearing potential, must have a negative pregnancy test
* Provide written informed consent

Exclusion Criteria:

* Clinically unstable patients, e.g., those who are clinically in decompensated heart failure or having active chest pain or presenting for admission with an unstable anginal syndrome
* Patients in whom introduction of a catheter into the left ventricle is contraindicated or would potentially be dangerous, e.g., patients with active ventricular arrhythmias or with significant aortic valve stenosis where crossing the aortic valve may be difficult and not clinically necessary
* Patients with anatomic right-to-left, bi-directional, or transient right-to-left cardiac shunts where Definity could traverse as a bolus
* Patients with known hypersensitivity to Definity
* Females who are pregnant or nursing

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Agreement between SHAPE and pressure catheter measurements | up to 1 day
  Correlation
Error between SHAPE and pressure catheter measurements | up to 1 day
  ANOVA/Post-hoc comparisons

CONTACTS AND LOCATIONS:
Overall Officials: Jaydev Dave, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University and Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will generate pressure values in the aorta, and left and right ventricles using the proposed research method (i.e., SHAPE) and using the standard of care (i.e., catheter based pressure values). Additionally peripheral and central pressures will be generated. All of the pressure values will be made available. Further, all ultrasound data obtained for SHAPE measurements will be made available after anonymizing the data-set to remove any patient information.
Supporting Information: ICF
Time Frame: 2019-05-30 (anticipated) or starting 6 months after publication
Access Criteria: Accessible research platform

REFERENCES:
- [Background] Dave JK, Halldorsdottir VG, Eisenbrey JR, Liu JB, McDonald ME, Dickie K, Leung C, Forsberg F. Noninvasive estimation of dynamic pressures in vitro and in vivo using the subharmonic response from microbubbles. IEEE Trans Ultrason Ferroelectr Freq Control. 2011 Oct;58(10):2056-66. doi: 10.1109/TUFFC.2011.2056. PMID 21989870
- [Background] Dave JK, Halldorsdottir VG, Eisenbrey JR, Forsberg F. Processing of subharmonic signals from ultrasound contrast agents to determine ambient pressures. Ultrason Imaging. 2012 Apr;34(2):81-92. doi: 10.1177/016173461203400202. PMID 22724314
- [Background] Dave JK, Halldorsdottir VG, Eisenbrey JR, Merton DA, Liu JB, Machado P, Zhao H, Park S, Dianis S, Chalek CL, Thomenius KE, Brown DB, Forsberg F. On the implementation of an automated acoustic output optimization algorithm for subharmonic aided pressure estimation. Ultrasonics. 2013 Apr;53(4):880-8. doi: 10.1016/j.ultras.2012.12.010. Epub 2013 Jan 2. PMID 23347593
- [Background] Dave JK, Halldorsdottir VG, Eisenbrey JR, Raichlen JS, Liu JB, McDonald ME, Dickie K, Wang S, Leung C, Forsberg F. Subharmonic microbubble emissions for noninvasively tracking right ventricular pressures. Am J Physiol Heart Circ Physiol. 2012 Jul;303(1):H126-32. doi: 10.1152/ajpheart.00560.2011. Epub 2012 May 4. PMID 22561300
- [Background] Dave JK, Halldorsdottir VG, Eisenbrey JR, Raichlen JS, Liu JB, McDonald ME, Dickie K, Wang S, Leung C, Forsberg F. Noninvasive LV pressure estimation using subharmonic emissions from microbubbles. JACC Cardiovasc Imaging. 2012 Jan;5(1):87-92. doi: 10.1016/j.jcmg.2011.08.017. PMID 22239898
- [Background] Eisenbrey JR, Dave JK, Halldorsdottir VG, Merton DA, Miller C, Gonzalez JM, Machado P, Park S, Dianis S, Chalek CL, Kim CE, Baliff JP, Thomenius KE, Brown DB, Navarro V, Forsberg F. Chronic liver disease: noninvasive subharmonic aided pressure estimation of hepatic venous pressure gradient. Radiology. 2013 Aug;268(2):581-8. doi: 10.1148/radiol.13121769. Epub 2013 Mar 22. PMID 23525208
- [Background] Forsberg F, Liu JB, Shi WT, Furuse J, Shimizu M, Goldberg BB. In vivo pressure estimation using subharmonic contrast microbubble signals: proof of concept. IEEE Trans Ultrason Ferroelectr Freq Control. 2005 Apr;52(4):581-3. doi: 10.1109/tuffc.2005.1428040. PMID 16060506
- [Background] Halldorsdottir VG, Dave JK, Leodore LM, Eisenbrey JR, Park S, Hall AL, Thomenius K, Forsberg F. Subharmonic contrast microbubble signals for noninvasive pressure estimation under static and dynamic flow conditions. Ultrason Imaging. 2011 Jul;33(3):153-64. doi: 10.1177/016173461103300301. PMID 21842580
- [Background] Shi WT, Forsberg F, Raichlen JS, Needleman L, Goldberg BB. Pressure dependence of subharmonic signals from contrast microbubbles. Ultrasound Med Biol. 1999 Feb;25(2):275-83. doi: 10.1016/s0301-5629(98)00163-x. PMID 10320317
- [Background] Halldorsdottir VG, Dave JK, Eisenbrey JR, Machado P, Zhao H, Liu JB, Merton DA, Forsberg F. Subharmonic aided pressure estimation for monitoring interstitial fluid pressure in tumours--in vitro and in vivo proof of concept. Ultrasonics. 2014 Sep;54(7):1938-44. doi: 10.1016/j.ultras.2014.04.022. Epub 2014 May 6. PMID 24856899
- [Derived] Esposito C, Machado P, McDonald ME, Savage MP, Fischman D, Mehrotra P, Cohen IS, Ruggiero N 2nd, Walinsky P, Vishnevsky A, Dickie K, Davis M, Forsberg F, Dave JK. Noninvasive Evaluation of Cardiac Chamber Pressures Using Subharmonic-Aided Pressure Estimation With Definity Microbubbles. JACC Cardiovasc Imaging. 2023 Feb;16(2):224-235. doi: 10.1016/j.jcmg.2022.09.013. Epub 2022 Nov 16. PMID 36648035
- [Derived] Esposito C, Machado P, Cohen IS, Mehrotra P, Savage M, Fischman D, Davis M, Ruggiero N, Walinsky P, McDonald ME, Dickie K, Forsberg F, Dave JK. Comparing Central Aortic Pressures Obtained Using a SphygmoCor Device to Pressures Obtained Using a Pressure Catheter. Am J Hypertens. 2022 May 10;35(5):397-406. doi: 10.1093/ajh/hpac010. PMID 35079778